CLINICAL TRIAL: NCT07280858
Title: A 2-Stage, Phase I/II, Active-controlled, Randomized, Observer-blinded, Dose-finding Study to Assess the Safety, Reactogenicity, and Immunogenicity of a Broadly Protective Sarbecovirus Vaccine (GBP511) in Healthy Adults (Aged 18 Years and Older)
Brief Title: A Phase I/II, Dose-finding Study to Assess the Safety, Reactogenicity, and Immunogenicity of a Broadly Protective Sarbecovirus Vaccine (GBP511) in Healthy Adults.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GBP511_001
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants; Sarbecovirus
MeSH Terms: interventions — BNT162 Vaccine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Stage 1: sequential, Stage 2 : parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Test Group 1-1 (GBP511) (Experimental): Low-dose of recombinant protein nanoparticle pan-Sarbecovirus vaccine (2µg of RBD/strain); a total injection volume of 0.5mL
  IM injections on Day 1, 29 (Visit 2, 5)
  Interventions: Biological: Test Drug 1-1 (GBP511 low dose)
- Test Group 1-2 (GBP511+CAS-1) (Experimental): Low-dose of recombinant protein nanoparticle pan-Sarbecovirus vaccine (2µg of RBD/strain) adjuvanted with a standard dose of CAS-1; a total injection volume of 0.5mL
  IM injections on Day 1, 29 (Visit 2, 5)
  Interventions: Biological: Test Drug 2-1 (GBP511 low dose + CAS-1)
- Control Group (Active Comparator): Comirnaty (2025-26 or subsequent seasonal formulation, 30 mcg of SARS-CoV-2 LP.8.1 spike protein mRNA); a total injection volume of 0.3mL Normal saline; a total injection volume of 0.5mL
  Comirnaty: IM injection on Day 1 (Visit 2) Normal Saline: IM injection on Day 29 (Visit 5)
  Interventions: Biological: Comparator (Comirnaty); Biological: Placebo (Normal Saline)
- Test group 1-3 (GBP511) (Experimental): Mid-dose of recombinant protein nanoparticle pan-Sarbecovirus vaccine (6µg of RBD/strain); a total injection volume of 0.5mL IM injections on Day 1, 29 (Visit 2, 5)
  Interventions: Biological: Test Drug 1-2 (GBP511 mid dose)
- Test group 1-4 (GBP511+CAS-1) (Experimental): Mid-dose of recombinant protein nanoparticle pan-Sarbecovirus vaccine (6µg of RBD/strain) adjuvanted with a standard dose of CAS-1; a total injection volume of 0.5mL IM injections on Day 1, 29 (Visit 2, 5)
  Interventions: Biological: Test Drug 2-2 (GBP511 mid dose + CAS-1)
- Test Group 1-5 (GBP511) (Experimental): High-dose of recombinant protein nanoparticle pan-Sarbecovirus vaccine (18µg of RBD/strain); a total injection volume of 0.5mL IM injections on Day 1, 29 (Visit 2, 5)
  Interventions: Biological: Test Drug 1-3 (GBP511 high dose)
- Test Group 1-6 (GBP511+CAS-1) (Experimental): High-dose of recombinant protein nanoparticle pan-Sarbecovirus vaccine (18µg of RBD/strain) adjuvanted with a standard dose of CAS-1; a total injection volume of 0.5mL IM injections on Day 1, 29 (Visit 2, 5)
  Interventions: Biological: Test Drug 2-3 (GBP511 high dose + CAS-1)
- Test Group 2-1 (Stage 2) (Experimental): Participants will receive 2 intramuscular injections of the test vaccine in stage 2.
  Injections on Day 1, 29 (Visit 2, 5), in line with the selected dose regimen in stage 1.
  Interventions: Biological: Test Drug 13 (Stage 2, GBP511-A or B)
- Test Group 2-2 (Stage 2) (Experimental): Participants will receive 2 intramuscular injections of the test vaccine in stage 2.
  Injections on Day 1, 29 (Visit 2, 5), in line with the selected dose regimen in stage 1.
  Interventions: Biological: Test Drug 14 (Stage 2, GBP511-A or B)

INTERVENTIONS:
Biological: Test Drug 1-1 (GBP511 low dose) — injection volume of 0.5mililiter (mL) with 2-doses at 4 weeks interval in stage 1 and 1-dose or 2-doses at 4 weeks interval in stage 2.
  Low dose: 2μg/strain, Mid dose: 6μg/strain, High dose: 18μg/strain
  Arms: Test Group 1-1 (GBP511)
Biological: Test Drug 1-2 (GBP511 mid dose) — injection volume of 0.5mililiter (mL) with 2-doses at 4 weeks interval in stage 1 and 1-dose or 2-doses at 4 weeks interval in stage 2.
  Low dose: 2μg/strain, Mid dose: 6μg/strain, High dose: 18μg/strain
  Arms: Test group 1-3 (GBP511)
Biological: Test Drug 1-3 (GBP511 high dose) — injection volume of 0.5mililiter (mL) with 2-doses at 4 weeks interval in stage 1 and 1-dose or 2-doses at 4 weeks interval in stage 2.
  Low dose: 2μg/strain, Mid dose: 6μg/strain, High dose: 18μg/strain
  Arms: Test Group 1-5 (GBP511)
Biological: Test Drug 2-1 (GBP511 low dose + CAS-1) — injection volume of 0.5mililiter (mL) with 2-doses at 4 weeks interval in stage 1 and 1-dose or 2-doses at 4 weeks interval in stage 2.
  GBP511 - Low dose: 2μg/strain, Mid dose: 6μg/strain, High dose: 18μg/strain CAS-1 standard adjuvant dose
  Arms: Test Group 1-2 (GBP511+CAS-1)
Biological: Test Drug 2-2 (GBP511 mid dose + CAS-1) — injection volume of 0.5mililiter (mL) with 2-doses at 4 weeks interval in stage 1 and 1-dose or 2-doses at 4 weeks interval in stage 2.
  GBP511 - Low dose: 2μg/strain, Mid dose: 6μg/strain, High dose: 18μg/strain CAS-1 standard adjuvant dose
  Arms: Test group 1-4 (GBP511+CAS-1)
Biological: Test Drug 2-3 (GBP511 high dose + CAS-1) — injection volume of 0.5mililiter (mL) with 2-doses at 4 weeks interval in stage 1 and 1-dose or 2-doses at 4 weeks interval in stage 2.
  GBP511 - Low dose: 2μg/strain, Mid dose: 6μg/strain, High dose: 18μg/strain CAS-1 standard adjuvant dose
  Arms: Test Group 1-6 (GBP511+CAS-1)
Biological: Comparator (Comirnaty) — injection volume of 0.3mililiter (mL) with single-dose at visit 2.
  30 mcg of SARS-CoV-2 LP.8.1 spike protein mRNA per 0.3mL
  Arms: Control Group
Biological: Placebo (Normal Saline) — injection volume of 0.5mililiter (mL) with single-dose at visit 5.
  Arms: Control Group
Biological: Test Drug 13 (Stage 2, GBP511-A or B) — Participants will receive 2 intramuscular injections of the test vaccine in stage 2.
  Injections on Day 1, 29 (Visit 2, 5), in line with the selected dose regimen in stage 1.
  Arms: Test Group 2-1 (Stage 2)
Biological: Test Drug 14 (Stage 2, GBP511-A or B) — Participants will receive 2 intramuscular injections of the test vaccine in stage 2.
  Injections on Day 1, 29 (Visit 2, 5), in line with the selected dose regimen in stage 1.
  Arms: Test Group 2-2 (Stage 2)

SUMMARY:
The purpose of this research study is to evaluate the safety of and the body's immune response to single and multiple vaccinations in healthy men and women. We want to find out what effects GBP511 has on you and your health. We are doing this study to find out:

If the study drug has any side effects when given as single and multiple vaccinations.

If reactogenicity, an indication that the immune systems is working and is preparing to protect the body against future infection, occurs. This is a normal physical inflammatory response that occurs after vaccination, manifesting as localised reactions that may include pain or redness at the injection site, or systemic symptoms such as headache or fever.

If immunogenicity which is when GBP511 causes your body to make antibodies against the non-harmful viral proteins contained within GBP511, called 'neutralising antibodies (Nab),' occurs. And if GBP511 will cause the specialised cells of the body's immune system to mount a defence against the non-harmful viral proteins contained within GBP511, called 'cell-mediated immunity (CMI)'.

In this study, GBP511 will be administered with and without adjuvant, CAS-1. An adjuvant is an ingredient used in some vaccines that help produce a stronger immune response in the people receiving the vaccine and thus helps the vaccine work better.

This study will recruit approximately 368 participants in total and will be conducted in two stages:

Stage 1 will look at two vaccinations with GBP511 when given with and without the CAS-1 adjuvant; and Stage 2 will look at either one or two vaccinations with two candidate GBP511 vaccines chosen from Stage 1 of the study.

Participants will be required to attend Linear's clinical unit on two separate occasions to receive their two vaccinations. On the first day of dosing (Visit 2/Day 1) and second day of dosing (Visit 5/Day 29), we will be testing a single dose of the study drug in up to 168 healthy volunteers who will be divided into 3 groups. Group 1, Groups 2 and 3 will have 56 people each. These 3 groups will be divided into treatment subgroups, with a total of 6 test subgroups and 3 control subgroups. In all groups, neither you or the study doctor will know what subgroup you are part of, and therefore what treatment (GBP511 or Comirnaty+ placebo) you will receive.

ELIGIBILITY:
Inclusion Criteria:

Age

1. For Stage 1, participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.

   For Stage 2, participant must be 18 years of age and older, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participants who are healthy as determined by medical evaluation including medical history, vital signs, physical examination, clinical laboratory tests, and medical judgement of the investigator.
3. Participants who are willing and able to attend all scheduled visits and comply with all study procedures.
4. Body mass index (BMI) within the range of 18.5-32.0 kg/m2 (revised) at screening
5. Participants who received a primary series and at least one booster dose of an authorized COVID-19 vaccine at least 24 weeks prior to the 1st study vaccination.

   Sex and Contraceptive/Barrier Requirements
6. All participants must agree to be abstinent from heterosexual intercourse or agree to consistently use at least one acceptable method of contraception from at least 4 weeks prior to the 1st study vaccination to 12 weeks after the last study vaccination (See Appendix 10.4 for detailed contraceptive methods).
7. Women of childbearing potential (WOCBP) with a negative urine or serum pregnancy test at screening.

   * Female participants who are surgically sterile (e.g., having undergone a full hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal with at least 12 months amenorrhoea not considered to be caused by any other medical condition, are not subject to a pregnancy test.

   Informed Consent
8. Participants who are capable of giving signed informed consent as described in Appendix 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol before initiation of any trial-specific procedures.

Exclusion Criteria:

Medical Conditions

1. Any clinically significant respiratory symptoms (e.g., cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 24 hours prior to the 1st study vaccination. Prospective participants with these conditions cannot be included until 24 hours after resolution.
2. Concurrent or a history of virologically or serologically confirmed SARS-CoV-2 infection, or suspected SARS-CoV-2 infection as determined by the investigator, within 24 weeks prior to the 1st study vaccination.
3. History of virologically or serologically confirmed SARS-CoV-1, or MERS disease.
4. History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease.
5. Any positive test results for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening.
6. History of bleeding disorder or thrombocytopenia which is contraindicating intramuscular vaccination in the investigator's opinion.
7. History of hypersensitivity and severe allergic reaction (e.g., anaphylaxis) to any vaccines or components of the study intervention.
8. History of neurologic diseases (e.g., Guillain-Barre syndrome, myelitis, or encephalomyelitis).
9. History of myocarditis, pericarditis or myopericarditis, as assessed by the investigator, indicating probable or possible myocarditis, pericarditis, or myopericarditis, or demonstrating clinically significant abnormalities that could affect participant safety or the interpretation of study findings.
10. History of malignancy within 1 year prior to first study vaccination, except for cutaneous non-melanoma malignancy, melanoma-in-situ, or cervical carcinoma in situ that have been fully treated with completed follow-up prior to screening. Malignancy considered to carry minimal risk of recurrence may also be permitted at the discretion of the investigator.
11. Significant unstable chronic or acute illness that, in the opinion of the investigator, might pose a health risk to the participant if enrolled, or could interfere with the protocol-specified activities, or interpretation of study results.
12. Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g., alcohol or drug abuse, neurologic or psychiatric conditions).
13. Female participants who are pregnant or breastfeeding.

    Prior/Concomitant therapy
14. Receipt of any COVID-19 vaccination including investigational vaccines within 24 weeks prior to the 1st study vaccination or planned receipt at any time during the study period.
15. Receipt of any vaccinations intended to prevent SARS-CoV-1 or MERS, including investigational vaccines.
16. Receipt of any vaccine within 4 weeks prior to the 1st study vaccination or planned receipt of any vaccine through 4 weeks after the last study vaccination, except for influenza vaccination, which may be received at least 2 weeks prior to the 1st study vaccination.
17. Receipt of any immunoglobulins and/or blood-derived products within 12 weeks prior to the 1st study vaccination or planned receipt at any time during the study period.
18. Receipt of immunosuppressive therapy, such as any use of anti-cancer chemotherapy or radiation therapy; or chronic use of systemic corticosteroid (≥10 mg prednisone/day or equivalent more than 14 consecutive days) within 12 weeks prior to the 1st study vaccination and throughout the entire study period. The use of intranasal, inhaled, topical, or intra-articular corticosteroid is permitted.

    Prior/Concurrent Clinical Study Experience
19. Participation in another clinical study and receipt of study intervention within 4 weeks prior to the 1st study vaccination, or concurrent, planned participation in another clinical study with study intervention during this study period.

    Other Exclusions
20. Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.
21. Donation of ≥450mL of blood product within 4 weeks prior to screening, or planned donation of blood product from enrollment through 12 weeks after the last study vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2028-09-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing any immediate reactions | 30 minutes (2 hours for sentinel participants) following each study vaccination
  For stage 1
Percentage of participants reporting any solicited local AEs | during the 7 days following each study vaccination
  For stage 1
Percentage of participants reporting any solicited systemic AEs | during the 7 days following each study vaccination
  For stage 1
Percentage of participants experiencing any unsolicited AEs | during the 28 days following each study vaccination
  For stage 1
Percentage of participants experiencing any SAEs, MAAEs, AESIs, as well as AE leading to study withdrawal | 1st Vaccination date, 1 week, 2 weeks, 4 weeks following the 1st study vaccination, and 2nd vaccination date, 1 week, 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For stage 1
GMT of neutralizing antibody against each matched strain measured by a pseudo-virus neutralization assay at each time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
  For stage 2
GMR of neutralizing antibody against each matched strain measured by a pseudo-virus neutralization assay, from each pre-vaccination to subsequent time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
  For stage 2
Percentage of participants with ≥ 2-fold and 4-fold rises against each matched strain in pseudo-virus neutralizing antibody titer, from baseline to each subsequent time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
  For stage 2

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of neutralizing antibody against each matched strain measured by a pseudo-virus neutralization assay | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For stage 1
Geometric mean ratio (GMR) of neutralizing antibody against each matched strain measured by a pseudo-virus neutralization assay | From pre-vaccination to baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For stage 1
Percentage of participants with ≥ 2-fold and 4-fold rises against each matched strain in pseudo-virus neutralizing antibody titer | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For stage 1
GMT of RBD-binding IgG antibody against each matched strain measured by ECL assay at each time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination (following the last vaccination for stage 2)
  For stage 1,2
GMR of RBD-binding IgG antibody against each matched strain measured by ECL assay, from each pre-vaccination to subsequent time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination(following the last vaccination for stage 2).
  For stage 1,2
Percentage of participants with ≥ 2-fold and 4-fold rises in RBD-binding IgG titer against each matched strain, measured by ECL assay, from baseline to each subsequent time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination(following the last vaccination for stage 2).
  For stage 1,2
GMT of neutralizing antibody against each mismatched strain measured by a pseudo-virus neutralization assay at each time point. | baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination (following the last vaccination for stage 2).
  For Stage 1, The endpoints will be evaluated exclusively in a subset of approximately 33% of participants at the following time points:
  baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For Stage 2, The endpoints will be evaluated exclusively in a subset of approximately 20% of participants at the following time points:
  baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
GMR of neutralizing antibody against each mismatched strain measured by a pseudo-virus neutralization assay, from each pre-vaccination to subsequent time point. | baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination (following the last vaccination for stage 2).
  For Stage 1, The endpoints will be evaluated exclusively in a subset of approximately 33% of participants at the following time points:
  baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For Stage 2, The endpoints will be evaluated exclusively in a subset of approximately 20% of participants at the following time points:
  baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
Percentage of participants with ≥ 2-fold and 4-fold rises against each mismatched strain in pseudo-virus neutralizing antibody titer, from baseline to each subsequent time point. | baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination (following the last vaccination for stage 2).
  For Stage 1, The endpoints will be evaluated exclusively in a subset of approximately 33% of participants at the following time points:
  baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For Stage 2, The endpoints will be evaluated exclusively in a subset of approximately 20% of participants at the following time points:
  baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
Cell-mediated response for both Th1 and Th2 cytokines (including but not limited to IFN-γ, IL-2, and IL-4 produced by T lymphocytes) measured by FluoroSpot | baseline, 2 weeks following the 1st study vaccination, and 2 weeks, and 6 months following the 2nd study vaccination(following the last vaccination for stage 2).
  For Stage 1, The following endpoint will be evaluated exclusively in sentinel participants at the following time points:
  baseline, 2 weeks following the 1st study vaccination, and 2 weeks, and 6 months following the 2nd study vaccination.
  For Stage 2, The following endpoints will be evaluated exclusively in a subset of approximately the first 20% of participants at the following time points:
  baseline, 2 weeks following the 1st study vaccination, and 2 weeks, and 6 months following the last study vaccination.
Percentage of participants experiencing any immediate reactions | within 30 minutes following each study vaccination
  For stage 2
Percentage of participants reporting any solicited local AEs | during the 7 days following each study vaccination
  For stage 2
Percentage of participants reporting any solicited systemic AEs | during the 7 days following each study vaccination
  For stage 2
Percentage of participants experiencing any unsolicited AEs | during the 28 days following each study vaccination
  For stage 2
Percentage of participants experiencing any SAEs, MAAEs, AESIs, as well as AE leading to study withdrawal | during the entire study period
  For stage 2

OTHER OUTCOMES:
GMT of neutralizing antibody against each strain measured by a pseudo-virus neutralization assay at each time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
  For Stage 1&2, some of the following endpoints may be evaluated in a subset of participants at all or partial time points.
GMR of neutralizing antibody against each strain measured by a pseudo-virus neutralization assay, from each pre-vaccination to subsequent time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
  For Stage 1&2, some of the following endpoints may be evaluated in a subset of participants at all or partial time points.
Percentage of participants with ≥ 2-fold and 4-fold rises against each strain in pseudo-virus neutralizing antibody titer, from baseline to each subsequent time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the last study vaccination.
  For stage 1& 2, Some of the following endpoints may be evaluated in a subset of participants at all or partial time points.
GMT ratios of neutralizing antibody against each matched and mismatched strain measured by a pseudo-virus neutralization assay | Vaccination date, 2 weeks, 4 weeks, 3 months, 6 months, 12 months following the vaccination date.
  For Stage 2
GMT ratios of RBD-binding IgG antibody against each matched strain measured by ECL | Vaccination date, 2 weeks, 4 weeks, 3 months, 6 months, 12 months following the vaccination date.
  For Stage 2
Further evaluation of the safety and/or immunogenicity of GBP511 candidates may also be conducted using samples collected from study participants to undertake a range of exploratory analyses. | - Stage 1 and Stage 2: 1st vaccination date, 2 weeks, 2nd vaccination date, 2 week, 4 week, 3 months, 6 month, 12 month - Stage 2 only: Vaccination date, 2 week, 4 week, 3 month, 6 month, 12 month
  For Stage 1&2

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Linear, Joondalup, Western Australia
  - Linear, Nedlands, Western Australia